CLINICAL TRIAL: NCT04722666
Title: A Double-blind, Placebo-controlled, Randomized Dose-ranging Trial to Investigate Efficacy and Safety of Intravenous MIJ821 Infusion in Addition to Comprehensive Standard of Care on the Rapid Reduction of Symptoms of Major Depressive Disorder in Subjects Who Have Suicidal Ideation With Intent
Brief Title: Study of Efficacy and Safety of MIJ821 in Addition to Comprehensive Standard of Care on the Rapid Reduction of Symptoms of Major Depressive Disorder in Subjects Who Have Suicidal Ideation With Intent
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated by Novartis
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMIJ821A12201
Record Dates: First submitted 2021-01-21; First posted 2021-01-25 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2023-10

CONDITIONS: Major Depressive Disorder With Suicidal Ideation With Intent
Keywords: Major Depressive Disorder; Mental disorder; Mood disorder; Depression; Suicide; Suicidal Ideation; Suicidal intent; Suicidal risk; Self-Injurious Behavior; MIJ821; Antidepressive Agent; Psychotropic Drug; Hospitalization; Intravenous; Placebo; Adult
MeSH Terms: conditions — Depressive Disorder, Major; Mental Disorders; Mood Disorders; Depression; Suicide; Suicidal Ideation; Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- MIJ821 (mg/kg) - very low dose (Experimental): MIJ821 (mg/kg) very low dose for 40 minutes IV infusion on Day 1, Day 15 and Day 29
  Interventions: Drug: MIJ821 Intravenous Injection
- MIJ821 (mg/kg) - low dose (Experimental): MIJ821 (mg/kg) low dose for 40 minutes IV infusion on Day 1, Day 15 and Day 29
  Interventions: Drug: MIJ821 Intravenous Injection
- MIJ821(mg/kg) - high dose (Experimental): MIJ821 (mg/kg) high dose for 40 minutes IV infusion on Day 1, Day 15 and Day 29
  Interventions: Drug: MIJ821 Intravenous Injection
- MIJ821 (mg/kg) - very high dose (Experimental): MIJ821 (mg/kg) very high dose for 40 minutes IV infusion on Day 1, Day 15 and Day 29
  Interventions: Drug: MIJ821 Intravenous Injection
- Placebo (Placebo Comparator): 40 minutes IV infusion of 0.9% sodium chloride on Day 1, Day 15 and Day 29
  Interventions: Drug: Placebo Intravenous Injection
- MIJ821 (mg/kg) - high dose/Placebo (Experimental): MIJ821 (mg/kg) high dose for 40 minutes IV infusion on Day 1/0.9% sodium chloride for 40 minutes IV infusion on Day 15 and Day 29
  Interventions: Drug: MIJ821 Intravenous Injection; Drug: Placebo Intravenous Injection
- MIJ821 (mg/kg) - very high dose/Placebo (Experimental): MIJ821 (mg/kg) very high dose for 40 minutes IV infusion on Day 1/0.9% sodium chloride for 40 minutes IV infusion on Day 15 and Day 29
  Interventions: Drug: MIJ821 Intravenous Injection; Drug: Placebo Intravenous Injection

INTERVENTIONS:
Drug: MIJ821 Intravenous Injection — MIJ821 supplied in vials to be prepared on a mg/kg basis and to be administered for 40 minutes IV infusion on Day 1, Day 15 and Day 29
  Arms: MIJ821 (mg/kg) - high dose/Placebo; MIJ821 (mg/kg) - low dose; MIJ821 (mg/kg) - very high dose; MIJ821 (mg/kg) - very high dose/Placebo; MIJ821 (mg/kg) - very low dose; MIJ821(mg/kg) - high dose
Drug: Placebo Intravenous Injection — 40 minutes IV infusion of 0.9% sodium chloride solution on Day1, Day 15 and Day 29
  Arms: MIJ821 (mg/kg) - high dose/Placebo; MIJ821 (mg/kg) - very high dose/Placebo; Placebo

SUMMARY:
Study of efficacy and safety of MIJ821 in addition to comprehensive standard of care on the rapid reduction of symptoms of Major Depressive Disorder (MDD) in subjects who have suicidal ideation with intent

DETAILED DESCRIPTION:
The main purpose of this study is to support the dose selection for future Phase III clinical trials by evaluating efficacy and safety of four MIJ821 doses (very low, low, high and very high) administered every other week by intravenous infusion on top of pharmacological antidepressant treatment, compared with placebo, for the rapid reduction of the symptoms of MDD in participants who have suicidal ideation with intent. In addition, the study will explore the effect of single dose administration of very high and high doses to treat MDD in participants who have suicidal ideation with intent.

The study consists of three periods: a Screening Period (up to 48 hrs), a double-blind Core Period (6 weeks) and Extension Period (up to 52 weeks). The Extension Period will explore durability of the effect of the study treatment and the effect of MIJ821 on relapse rate, as well as safety of repeated MIJ821 administration.

All patients in the extension period will receive active treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the study
2. Male and female participants, 18 to 65 years of age (inclusive) at screening
3. DSM-5 defined major depressive disorder (MDD) with a current major depressive episode (MDE) without psychotic features at the time of screening based upon clinical assessment and confirmed by the Mini International Neuropsychiatric Interview (M.I.N.I.) assessed at Screening
4. Participants must have current suicidal ideation with intent, confirmed by a "Yes" response to Question B3 AND either Question B10 or Question B11 obtained from the M.I.N.I., assessed at Screening
5. Current suicidal ideation with intent, confirmed by "Yes" response to Question 3 AND either Question 9 or Question 10 obtained from the SSTS at Baseline
6. Montgomery-Åsberg Depression Rating Scale (MADRS) score > 28 at Screening and before randomization on Day 1
7. Participants must agree to receive pharmacological standard of care treatment to treat their MDD (as determined by the treating physician(s) based on clinical judgement and local treatment guidelines) during the trial duration
8. In the physician's opinion, acute psychiatric hospitalization is clinically warranted to treat the patient's condition, and the patient is either already in the hospital or agrees to be hospitalized voluntarily for the required per protocol period

Exclusion Criteria:

1. Any prior or current diagnosis of bipolar disorder, MDD with psychotic features, schizophrenia, or schizoaffective disorder as obtained from M.I.N.I. at Screening
2. Patients with acute alcohol or substance use disorder or withdrawal symptoms requiring detoxification, or patients who went through detoxification treatment (inpatient or outpatient) within 1 month before Screening.
3. Participant has a current clinical diagnosis of autism, dementia, or intellectual disability
4. History of seizures. Note: childhood febrile seizures are not exclusionary
5. Participants with borderline personality disorder as obtained from M.I.N.I. at Screening.
6. Participants with suicidal ideation or behavior caused primarily by another non-MDD condition as obtained from M.I.N.I. at Screening
7. Participants taking medications prohibited by the protocol
8. Intake of the following medications/ psychotherapy:

   1. Esketamine or Ketamine 2 months before Screening
   2. Monoamine oxidase inhibitors (MAOIs) 14 days before Screening
   3. Non-stable psychotherapy regimen and/or started less than 6 weeks before Screening
9. Any other condition (e.g. known liver disease/liver dysfunction, active malignancy, etc.) which in the opinion of the investigator would put the safety of the participant at risk, impede compliance or hinder completion of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the total score of the Montgomery Åsberg Depression Rating Scale (MADRS) | Baseline (first infusion) at 24 hours and up to 52 weeks
  The Montgomery Åsberg Depression Rating Scale (MADRS, SIGMA version), is a clinician rated scale designed to measure depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition. The MADRS evaluates apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts and suicidal thoughts. The MADRS will be collected electronically by qualified personnel

SECONDARY OUTCOMES:
Number and severity of treatment-emergent adverse events (TEAEs) and adverse events of special interest (AESI) | Baseline up to 6 weeks
  Treatment-emergent adverse events (TEAEs) and adverse events of special interest (AESIs) will be collected at all study visits
Pharmacokinetics (PK) of MIJ821 in plasma | Baseline up to 52 weeks
  PK parameters of MIJ821 in plasma after 1st infusion described by AUClast, Cmax, Tmax and after each other infusion described by Cmax and Tmax. In order to better define the PK profile, the timing of the PK sample collection may be altered based on emergent data.
Percentage of participants meeting response criteria of ≥50% reduction | Baseline up to 6 weeks
  Response criteria of ≥50% reduction from baseline in MADRS total score over time in the Core Period.
Percentage of participants meeting criteria for sustained response of ≥50% reduction | Baseline up to 6 weeks
  Sustained response from baseline in MADRS total score for a period of at least four weeks in the Core Period
Percentage of participants meeting remission criteria of MADRS total score of ≤12 | Baseline up to 6 weeks
  Remission criteria of MADRS total score of ≤12 over time in the Core Period
Percentage of participants meeting sustained remission criteria of MADRS total score of ≤12 | Baseline up to 6 weeks
  Remission criteria of MADRS total score of ≤12 sustained for a period of at least four weeks in the Core Period
Percentage of participants meeting criteria for relapse in the Extension Period | From 6 weeks up to 52 weeks
  Relapse for all patients meeting criteria for relapse over fixed period in the Extension Period
Percentage of relapsing participants meeting response criteria or remission criteria after the first infusion | From 6 weeks up to 52 weeks
  Relapsing participants meeting response criteria or remission criteria after the first infusion of MIJ821 retreatment in the Extension Period

CONTACTS AND LOCATIONS:
Locations (35):
- United States (6):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Farmington, Connecticut
  - Novartis Investigative Site, Oakland Park, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Rockville, Maryland
  - Novartis Investigative Site, DeSoto, Texas
- Novartis Investigative Site, Buenos Aires, Argentina
- Brazil (2):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, São Bernardo do Campo, São Paulo
- Novartis Investigative Site, Toronto, Ontario, Canada
- Germany (2):
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, München
- Japan (3):
  - Novartis Investigative Site, Toyoake, Aichi-ken
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Kodaira, Tokyo
- Malaysia (2):
  - Novartis Investigative Site, Seremban, Negeri Sembilan
  - Novartis Investigative Site, Kuala Lumpur
- Mexico (3):
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, Mazatlán, Sinaloa
  - Novartis Investigative Site, San Luis Potosí City
- Novartis Investigative Site, Groningen, Netherlands
- Poland (5):
  - Novartis Investigative Site, Pruszków, Masovian Voivodeship
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Swiecie n/W
  - Novartis Investigative Site, Lodz, Łódź Voivodeship
- Novartis Investigative Site, Moscow, Russia
- Spain (4):
  - Novartis Investigative Site, Palma de Mallorca, Balearic Islands
  - Novartis Investigative Site, Vitoria-Gasteiz, Basque Country
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Barcelona
- Novartis Investigative Site, Taipei, Taiwan
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Bursa, Gorukle
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Izmir

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/